CLINICAL TRIAL: NCT02471560
Title: The Effect of Tecfidera® (Dimethyl Fumarate, BG00012) on the Gut Microbiota as a Causal Factor for Gastro Intestinal Associated Adverse Events.
Brief Title: Tecfidera and the Gut Microbiota
Acronym: TECONGUT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NOR-BGT-14-10665; 2015-001197-18 (EudraCT Number)
Record Dates: First submitted 2015-06-11; First posted 2015-06-15 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Microbiota; DMF; Gastro intestinal; MS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Dimethyl Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dimethyl fumarate (Experimental): As prescribed by the Investigator according to the local Summary of Product Characteristics.
  Interventions: Drug: dimethyl fumarate
- injectable MS DMT (Active Comparator): As prescribed by the Investigator according to the local Summary of Product Characteristics.
  Interventions: Drug: injectable MS DMT

INTERVENTIONS:
Drug: dimethyl fumarate — As per the prevailing local label.
  Other Names: DMF; Tecfidera; BG00012
  Arms: dimethyl fumarate
Drug: injectable MS DMT — As described above.
  Arms: injectable MS DMT

SUMMARY:
The primary objective of the study is to determine if dimethyl fumarate (DMF) causes changes in the abundance and diversity of commensal microbiota. The secondary objectives of this study are as follows: To identify if there are differences in the gut microbiota composition between patients that do or do not develop gastro intestinal (GI) adverse events (AEs), both pre- and post DMF treatment and to examine if the resolution of GI AEs in DMF treated patients is reflected in the gut microbiota.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a confirmed diagnosis of RRMS and satisfy the therapeutic indication as described in the local label.
* Female subjects of childbearing potential who are not surgically sterile must practice effective contraception according to the summary of product characteristics (SPC) during their participation in the study and be willing and able to continue contraception for 30 days after their last dose of study treatment.

Key Exclusion Criteria:

* Diagnosis of primary progressive, secondary progressive or progressive relapsing MS.
* Antibiotic treatment in the last month prior to study entry.
* Scheduled alteration of diet, including the use of probiotics.

NOTE: Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-11-06 (Actual); Primary Completion 2017-06-12 (Actual); Study Completion 2017-06-12 (Actual)

PRIMARY OUTCOMES:
Comparison of the change in gut microbiota composition in participants pre vs. post initiation of DMF treatment. | Day 1, Week 2, Week 12 and/or upon occurrence of GI symptoms outside of designated time points

SECONDARY OUTCOMES:
Change in gut microbiota composition between DMF treated participants that do or do not develop GI AEs as measured by an increase in the Gastrointestinal Symptom Rating Scale (GSRS) score. | Day 1, Week 2, Week 12 and/or upon occurrence of GI symptoms outside of designated time points
  GSRS is a self-reported questionnaire regarding GI symptoms comprising 15 items scored on a 7-point Likert scale. The 15 items can be grouped in 5 dimensions 1) abdominal pain (abdominal pain, gastric hunger pain, and nausea) 2) reflux (heartburn and acid regurgitation) 3) indigestion (borborygmus, bloating, eructation, and increased flatus) 4) diarrhea (diarrhea, loose stools, and urgency) and 5) constipation (constipation, hard stools, incomplete evacuation). A GI AE will be defined as an at least 2 point (>=2) increase from baseline in total score of any of the 5 dimensions in the GSRS.
Changes in gut microbiota composition in participants treated with DMF compared to participants treated with an alternative injectable multiple sclerosis (MS) disease modifying therapies (DMT) | Day 1, Week 2, Week 12 and/or upon occurrence of GI symptoms outside of designated time points
Baseline differences in the gut microbiota composition between DMF treated participants that do or do not develop GI AEs. | Day 1, Week 2, Week 12 and/or upon occurrence of GI symptoms outside of designated time points
Changes in the gut microbiota composition of DMF treated participants after resolution of GI AEs vs. during GI AE occurrences. | Upon GI symptoms and week 12

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (7):
- Norway (7):
  - Research site, Drammen
  - Research site, Haukeland
  - Research Site, Lillehammer
  - Research site, Lørenskog
  - Research site, Molde
  - Research site, Oslo
  - Research site, Stavanger